CLINICAL TRIAL: NCT01439672
Title: Insulin Sensitivity, Impaired Counterregulation, and Glucose Variability
Acronym: BPK005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sue Brown, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15131; R01DK085623 (NIH)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Sensitivity (Experimental): Single arm. Each subject will consume a mixed meal beverage along with insulin administration in order to calculate insulin sensitivity.
  Interventions: Dietary Supplement: Mixed meal and insulin challenge

INTERVENTIONS:
Dietary Supplement: Mixed meal and insulin challenge — The subject will undergo a mixed meal and insulin challenge as follows: an insulin bolus will be administered and a mixed meal nutrition drink will be consumed over 1-5 minutes. The mixed meal nutrition drink will be selected for that individual to be most likely to raise the glucose levels by 100mg/dl and then return to baseline within a four-hour time period. The nutrition drink will selected from the following types of product lines: Boost products (Nestle Nutrition), Ensure products (Abbott Nutrition), Carnation Instant Breakfast (Nestle Nutrition) or Glucerna (Abbott Nutrition).The pre-meal insulin bolus will be calculated to bring the subject to ~100mg/dl at 1100.

SUMMARY:
This protocol will investigate physiological parameters including insulin sensitivity and counterregulatory function using a mixed meal test and induced hypoglycemia in subjects with type I diabetes.

DETAILED DESCRIPTION:
The principal idea of the proposed research is: in order to be successful, closed-loop control of glucose in diabetes must adapt to individual physiologic characteristics and to the behavioral profile of each person. We propose to build a system that will use observers of patients' behavior and metabolic state and control modules that are responsible for insulin delivery and hypoglycemia prevention. In this phase of the project, we will investigate relationships of insulin sensitivity and impaired counterregulation with blood glucose variability, aiming to develop algorithmic physiology observers, which will track specific parameters of glucose variability and recurrent hypoglycemia as markers of change in a person's insulin sensitivity and counterregulatory ability.

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetes mellitus (TIDM) (as defined by the American Diabetes Association criteria or judgment of a physician) for at least two years prior to the enrollment in the study.
* Use of an insulin pump to treat their diabetes for at least six months prior to the study.
* Ability to use a bolus calculator function with the current insulin pump with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor.
* Age 21 - 64 years. Adults age 65 and over are likely to have medical exclusions for the follow-up Phase 2 study, which involves induced hypoglycemia.
* Completed Phase 1 of the Institutional Review Board (IRB) #14956 "Development of a Behavioral Observer for Type 1 Diabetes Mellitus"
* Willingness to use lispro (Humalog) insulin two days prior to and during inpatient admission.
* Willingness to perform Self-Monitoring Blood Glucose (SMBG) 4 times per day at times before meals and bedtime.
* Demonstration of proper mental status and cognition for completion of the study.

Exclusion Criteria:

* Pregnancy
* Psychiatric disorders that would interfere with study tasks (e.g. mental retardation, substance abuse)
* History of a systemic deep tissue infection with methicillin-resistant staph aureus or Candida albicans
* Known bleeding diathesis or dyscrasia
* Active enrollment in another clinical trial
* Medical condition that would make operating an insulin pump difficult (e.g. blindness, severe arthritis, extensive scar tissue at sites where devices are inserted).
* Anemia (hematocrit <36% [females], <38% [males]),
* Allergy or adverse reaction to lispro (Humalog) insulin
* Conditions which may increase the risk of induced hypoglycemia such as symptomatic heart disease, congestive heart failure, history of a cerebrovascular event, atrial fibrillation, renal insufficiency (creatinine >1.5) or uncontrolled hypertension (resting blood pressure >140/90).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Center for Diabetes Technology, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Sensitivity
Started | 35
Completed | 11
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Sensitivity
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Measure insulin sensitivity following a mixed meal across admissions. Insulin sensitivity was measured based on the minimal model of glucose kinetics using plasma glucose and insulin obtained frequently (approximately every 5-15 minutes) in response to mixed meal challenge.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: 1/min per uU/mL
Groups:
- Insulin Sensitivity: Single arm. Each subject will consume a mixed meal beverage along with insulin administration in order to calculate insulin sensitivity. Each subject will be admitted twice approximately 3 weeks apart.
  Mixed meal and insulin challenge: The subject will undergo a mixed meal and insulin challenge as follows: an insulin bolus will be administered and a mixed meal nutrition drink will be consumed over 1-5 minutes. The mixed meal nutrition drink will be selected for that individual to be most likely to raise the glucose levels by 100mg/dl and then return to baseline within a four-hour time period. The nutrition drink will selected from the following types of product lines: Boost products (Nestle Nutrition), Ensure products (Abbott Nutrition), Carnation Instant Breakfast (Nestle Nutrition) or Glucerna (Abbott Nutrition).The pre-meal insulin bolus will be calculated to bring the subject to ~100mg/dl at 1100.
Arm/Group | Insulin Sensitivity
Number analyzed (Participants) | 11
1/min per uU/mL | 3.37*10^-4 (1.18*10^-4)

ADVERSE EVENTS:
Arm/Group | Insulin Sensitivity
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 2/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Sensitivity (N=35)
Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes